CLINICAL TRIAL: NCT06822049
Title: Improving Efficiency, Quality, and Equity: Randomized Controlled Evaluations of Remote vs. In-Person Clinical Trial Methods; Remote vs. In-Person Study Evaluation (RISE) Trials
Brief Title: Remote vs. In-Person Study Evaluation (RISE) Trials: RISE Above Smoking (Trial 1)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Collaborators: Medical University of South Carolina (Other); University of Pennsylvania (Other); University of Alabama at Birmingham (Other); National Center for Advancing Translational Sciences (NCATS) (NIH); Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Larry Hawk, Ph.D., professor, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STUDY00008797 (SUNY-Buff IRB); 1UG3TR004797-01A1 (NIH)
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-10

CONDITIONS: Remote vs. In-Person; Remote Visits; In-person Visits
Keywords: Remote vs. In-Person methods
MeSH Terms: interventions — Transdermal Patch

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group design.
  The study employs a two-stage adaptive biased-coin randomization technique. The initial randomization will be generated using a stratified biased coin design with an allocation probability of 0.75 and a randomization list within each stratum will be generated for both Stage I (randomization to remote vs in-person Intake) and Stage II (randomization to remote vs. in-person Treatment/Assessment visits). To optimize the balance in cell sizes across the 4 treatment conditions, the allocation probabilities will be adjusted at 3 study milestones (once 25%, 50%, and 75% of the target sample of 200 participants attend Treatment/Assessment Visit 1). Specifically, the allocation probability will be modified based on the imbalance in the number of participants across conditions who have attended Treatment/Assessment Visit 1.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- REMOTE intake AND REMOTE treatment/assessment (Other): In this arm, ppts have been randomly assigned to a REMOTE INTAKE eligibility/baseline visit, and subsequently randomized to 5 REMOTE treatment/assessment visits.
  Interventions: Drug: Combination Nicotine Replacement Therapy (patch and lozenge)
- REMOTE intake BUT IN-PERSON treatment/assessment (Other): In this arm, ppts have been randomly assigned to a REMOTE INTAKE eligibility/baseline visit, and subsequently randomized to 5 IN-PERSON treatment/assessment visits.
  Interventions: Drug: Combination Nicotine Replacement Therapy (patch and lozenge)
- IN-PERSON intake, BUT REMOTE treatment/assessment (Other): In this arm, ppts have been randomly assigned to an IN-PERSON INTAKE eligibility/baseline visit, and subsequently randomized to 5 REMOTE treatment/assessment visits.
  Interventions: Drug: Combination Nicotine Replacement Therapy (patch and lozenge)
- IN-PERSON intake AND IN-PERSON treatment/assessment (Other): In this arm, ppts have been randomly assigned to an IN-PERSON INTAKE eligibility/baseline visit, and subsequently randomized to 5 IN-PERSON treatment/assessment visits.
  Interventions: Drug: Combination Nicotine Replacement Therapy (patch and lozenge)

INTERVENTIONS:
Drug: Combination Nicotine Replacement Therapy (patch and lozenge) — All participants receive 8 weeks of combination nicotine replacement therapy - long-acting transdermal patch and short-acting lozenge.

SUMMARY:
The study will employ a randomized, parallel-group design with two-stage randomization. After an initial brief screen for basic eligibility, participants will be randomized (within site) to either Remote (R) or In-Person (IP) Intake Groups. During the Intake, detailed consent and eligibility assessment will be completed. Participants who are eligible at the Intake will be randomized (within site and Intake Group) to R or IP Treatment and Assessment Groups. Participants will be followed for 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Common to all 3 RCTs:

Inclusion criteria:

1. age18+ years
2. stable mailing address (for mailing study packets if assigned to Remote Intake and/or Remote Treatment/Assessment) within accessible range (1.5 hours) of each study site (per self report)
3. able to read, speak & verbally comprehend English
4. own an iOS or Android smartphone
5. have a valid e-mail address that is checked regularly or have regular access to text messages (to access follow-up assessments)

Specific to RCT 1:

Inclusion criteria:

a) daily cigarette smoker of 5+ cigarettes/day for 6+ months b) moderate or greater motivation to quit smoking (6+ on the Motivation to Stop Smoking Scale) d) agree to refrain from use of other tobacco products and use of non-study cessation treatments while participating in the trial e) Willing to be randomized to attend remote/in-person visits

Exclusion Criteria:

* Specific to RCT 1:

  a) use of tobacco/nicotine products other than cigarettes (except blunts, spliffs, cigars, little cigars, cigarillos) for average of 5_ days per week over the past 3 months b) prior allergy/intolerance to NRT patch or lozenge c). pregnant, breastfeeding, or planning to become pregnant in next 4 months d) use of varenicline, NRT (e.g., patch, gum, lozenge), or bupropion in past 7 days for purpose of quitting smoking e) consumption of >28 alcohol-containing drinks per week g) high risk involvement with illicit or nonmedical prescription drugs (NIDA-modified ASSIST=27+) h) suicide attempt with at least some wish to die in past 3 months i) mental illness (such as schizophrenia, bipolar disorder, or major depression) that led to hospitalization in the past 30 days j) unable/unwilling to provide informed consent or follow directions, inappropriately responsive, based on staff observations k) for participants age 21+: refusal to provide/show a pack of cigarettes for documentation at the intake visit

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Accrual efficiency/Pre-treatment visits | ~1 month
  Calculated from visit milestones. Of participants who were eligible on the Brief Screen, the percentage who who attend the (Remote vs. In-Person) Intake Visit, a major accrual bottleneck for in-person trials. Although pre-treatment participant loss from Intake to Clinic 1 is typically modest, we will also explore Intake to T/A Visit 1 (first dose of treatment) attrition and overall pre-treatment attrition (from Brief Screen to T/A Visit 1) for each group.
Trial Quality: Retention | ~3 months
  Retention will be assessed using visit milestone data to determine whether each participant achieved each T/A Visit (Visits 2-5) following T/A initiation at T/A Visit 1. We will calculate a continuous metric of retention (0-4; the number of visits completed) for each participant, supplemented by visit-specific data to provide a detailed examination of the time course and overall amount of retention.
Trial Quality: Treatment adherence/utilization (patient-reported) | 8 weeks (assessed at T/A Visits 3, 4, and 5)
  As in most studies in the smoking cessation clinical trial literature, we will assess self-reported patch and lozenge use since the previous visit and convert the data to percent adherence separately for patches and lozenges. Pharmacotherapy is initiated at T/A Visit 2; therefore treatment adherence is assessed at T/A Visits 3, 4, and 5).
Trial quality: Biospecimen completion rates | 3 months (assessed at T/A Visits 1,2, 3, 4, and 5)
  The number of visits (out of 5; T/A Visits 1-5) for which the biospecimen (expired-air CO) is obtained by the clinical site.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University at Buffalo, Buffalo, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
We plan to make available the full de-identified data set with metadata through the NAHDAP, a NIDA-funded platform for data sharing/archiving, with a topical focus on behavioral health data. NAHDAP operates under the umbrella of the ICPSR, based at the University of Michigan. Per the ICPSR website, the ICPSR is "the largest social science data archive in the world".
Supporting Information: Study Protocol, ICF
Time Frame: Consistent with NIH and Institute of Medicine recommendations, the data will be deposited no later than the publication of the primary study data or one year after each RCTs completion, whichever comes first. There is no planned end date.
Access Criteria: Data submitted for archiving/sharing will be consistent with Inter-university Consortium for Political and Social Research (ICPSR) and the National Addiction and HIV Data Archive Program (NAHDAP) data standards and data stewardship policies and will contain no personal identifiers. Typically, the data are publicly available via a unique digital object identifier (DOI).